CLINICAL TRIAL: NCT03586414
Title: Mitochondrial Targeted Antioxidant Supplementation and Diastolic Function in Healthy Men and Women
Brief Title: MitoQ Supplementation and Cardiovascular Function in Healthy Men and Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado Nutrition Obesity Research Center (NORC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-1782
Record Dates: First submitted 2018-02-21; First posted 2018-07-13 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diastolic Dysfunction
Keywords: MitoQ
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: 'MITOQUINOL MESYLATE then placebo (Experimental): 'MITOQUINOL MESYLATE' administered twice daily for 4 weeks followed by a washout, then placebo capsule administered twice daily for 4 weeks. Capsules with active product contain 20 mg of 'MITOQUINOL MESYLATE'.
  Interventions: Dietary Supplement: MITOQUINOL MESYLATE then placebo
- B: Placebo then 'MITOQUINOL MESYLATE' (Experimental): Placebo capsule administered twice daily for 4 weeks followed by a washout period, then 'MITOQUINOL MESYLATE' administered twice daily for 4 weeks. Capsules with active product contain 20 mg of 'MITOQUINOL MESYLATE'
  Interventions: Dietary Supplement: Placebo, then MITOQUINOL MESYLATE

INTERVENTIONS:
Dietary Supplement: MITOQUINOL MESYLATE then placebo — MITOQUINOL MESYLATE then placebo: 'MITOQUINOL MESYLATE' administered twice daily for 4 weeks followed by a washout, then placebo capsule administered twice daily for 4 weeks. Capsules with active product contain 20 mg of 'MITOQUINOL MESYLATE'.
  Other Names: MitoQ, Mitoquinol methanesulfonate
  Arms: A: 'MITOQUINOL MESYLATE then placebo
Dietary Supplement: Placebo, then MITOQUINOL MESYLATE — 'Placebo, then MITOQUINOL MESYLATE' : Placebo administered twice daily for 4 weeks followed by a washout, then 'MITOQUINOL MESYLATE' capsule administered twice daily for 4 weeks. Capsules with active product contain 20 mg of 'MITOQUINOL MESYLATE'.
  Other Names: MitoQ, Mitoquinol methanesulfonate
  Arms: B: Placebo then 'MITOQUINOL MESYLATE'

SUMMARY:
In this pilot study, the investigators will determine whether supplementation with a mitochondrial-targeted antioxidant (Mitoquinone (MitoQ)) improves mitochondrial function, left ventricular diastolic and vascular function.

DETAILED DESCRIPTION:
Heart failure affects over 5 million American adults and the risk of heart failure increases with age. Diastolic function typically declines with age. Targeting age-related causal factors leading to the decline in diastolic function in both women and men is a major public health initiative. In this pilot study, the investigators will determine whether supplementation with a mitochondrial-targeted antioxidant (Mitoquinone (MitoQ)) improves mitochondrial function, left ventricular diastolic and vascular function in older adults. As an exploratory aim, the investigators will determine whether there are differences between men and women in response to this supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. 50 - 75 years of age
2. sedentary-to-recreationally active (<3 days of vigorous exercise);
3. nonsmokers;
4. healthy, as determined by medical history, physical examination, standard blood chemistries.

Exclusion Criteria:

1. history of cancer
2. history of cardiovascular disease
3. unwilling or unable to take MitoQ supplement;
4. taking antioxidant vitamins, corticosteroids, or anti-inflammatory medications (e.g., aspirin);
5. taking sex hormone therapy
6. presence of menses within last 1 year;
7. taking any other medications (e.g., antihypertensives, lipid lowering medications) that would interact with MitoQ or impact CV function

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Changes in diastolic function | Baseline and 4 weeks
  Echocardiographic measurements of LV function (and structure) will be assessed; primary outcomes include peak early (E) to late (A) mitral inflow velocity ratio and E to peak early (e') mitral annular velocity ratio.

SECONDARY OUTCOMES:
Changes in arterial stiffness | Baseline and 4 weeks
  Parameters of arterial stiffness will be measured using SphygmoCor XCEL (Atcor) system (pulse-wave velocity [PWV], pulse wave analyses [PWA]).
Changes in brachial artery flow-mediated dilation | Baseline and 4 weeks
  Brachial artery diameter and flow velocity will be acquired and analyzed using Vascular Analysis Tools 5.5.1
Changes in endothelial function | Baseline and 4 weeks
  Measure parameters using digital peripheral arterial tonometry (Endo-PAT 2000)
Changes in arterial vascular coupling | Baseline and 4 weeks
  Measure ratio between arterial stiffness [Ea] and ventricular stiffness [ELv] estimated from echocardiographic measures.
Changes in mitochondrial function | Baseline and 4 weeks
  Measure parameters of mitochondrial respiration using high-resolution respirometry performed on permeabilized PBMCs (Oroboros Oxygraph O2k); perform venous endothelial cell mitochondrial protein analyses (Fusion, Fission proteins, SIRT1, mitoSox, MnSOD) and oxidative stress (nitrotyrosine, NADPHoxidase).

CONTACTS AND LOCATIONS:
Overall Officials: Shauna Runchey, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Pending